CLINICAL TRIAL: NCT06811103
Title: DEterminants of Decisional Autonomy In Chronic Pain Patients and Assessment of Treatment Effectiveness
Acronym: DEDICATE
Status: Recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DEDICATE
Record Dates: First submitted 2025-01-30; First posted 2025-02-06 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: patient reported outcome — after enrollment, patient will have to answer to several patient reported outcome (PRO) to evaluate their pain, and well being. They will also answer to the MacCatT PRO to assess their understanding, reasoning, appreciation and choice expression

SUMMARY:
Chronic pain is defined as an unpleasant sensory and emotional experience that persists for three months or more, affecting 20-30% of the global adult population. It can arise from primary conditions or as a consequence of diseases and is a significant source of disability. Chronic pain is no longer merely a symptom but often a disease itself, with neurological and psychosocial mechanisms. The biopsychosocial model introduced by George Engel in 1977 helps to consider the biological, psychological, social, and societal dimensions of chronic pain. Patients with chronic pain must adapt to new circumstances, acquiring new knowledge and coping skills to reach a new homeostasis. The goal is not necessarily pain elimination but enabling patients to manage their pain and continue daily activities effectively.

International guidelines suggest a patient-centered, interdisciplinary approach to managing chronic pain, with an emphasis on empowering patients, motivating them, and involving them in decision-making. Autonomy in decision-making is crucial in this context, encompassing both negative freedom (absence of external constraints) and positive freedom (the ability to make choices and realize one's potential). However, chronic pain can limit cognitive and functional abilities, potentially impeding a patient's autonomy. Research indicates that a significant proportion of chronic pain patients experience a deficit in decision-making autonomy.

This mixed-methods study aims to explore the determinants of decision-making autonomy in chronic pain patients and its impact on their treatment. Using the MacCAT-T assessment tool, which evaluates understanding, reasoning, appreciation, and choice expression, the study will examine the relationship between patients' autonomy levels and their health outcomes. The study will also assess how clinicians perceive patients' autonomy compared to the tool's findings.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient attending their first consultation for chronic pain between 01/01/2025 and 31/12/2025
* Francophone patient
* Patient capable of expressing their non-opposition to participation

Exclusion Criteria:

* Patient with significant visual or hearing impairment
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under judicial protection Patient who opposes the use of their data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient attending their first consultation for chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
influences on decision making (MacCAT-T) | enrollment
  The primary objective is to identify the socio-demographic, cognitive, educational, and medical factors that influence overall decision-making autonomy in chronic pain patients who are seeking treatment for the first time as assessed with the MacArthur Competence Assessment Tool-Treatment (MacCAT-T)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Paris Saint Joseph, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No